CLINICAL TRIAL: NCT04533087
Title: ImPACt on Invasive Fungal Infections by Immune Checkpoint Inhibition
Acronym: PACIFIC
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Sibylle C Mellinghoff, Resident physician and research affiliate, University of Cologne
Other Study IDs: PACIFIC
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Invasive Fungal Infections
Keywords: immune checkpoint; invasive fungal infection
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood and biopsy (e.g. BAL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Candida blood stream infection
  Interventions: Other: No intervention
- Aspergillosis
  Interventions: Other: No intervention
- Rare mold infections
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This observational study aims to compare immune checkpoint expression in blood samples from patients with invasive fungal infections (IFI) against healthy controls.

DETAILED DESCRIPTION:
Participating sites will screen patients with invasive aspergillosis for eligibility. The investigators will enroll patients with aspergillosis and healthy controls. Patients will be informed by study personnel. Samples for imune phenotyping will be obtained within 7 days after diagnosis of IFI. A bronchoalveolar lavage (BAL) biopsy is taken at initial diagnostic bronchoscopy or other biopsy during surgical debridement whenever applicable and feasible.

The following data items will be collected: Patient characteristics, details on invasive fungal infection (IFI), underlying disease, outcome after 90 days (response, remission, progress, death). All collected data will be interpreted at the end of the study. All patients must agree to participate and sign the informed consent form.

The primary objective is to compare immune checkpoint expression in blood samples from patients with IFI against healthy controls. Exploratively, lymphocytic immune phenotypes in BAL or other biopsy samples from patients with IFI will be assessed. Further, cytotoxic T cell responses in blood samples from patients with IFI shall be investigated and the level of immune checkpoint expression correlated with mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Proven or probable, incl. PCR, positive IFI along 2019 EORTC/MSG criteria
* Signed ICF

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with IFI and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Measurement of immune checkpoint expression levels in blood samples from patients with IFI and healthy controls by flowcytometry | 3 years
  To compare immune checkpoint expression in blood samples from patients with IFI against healthy controls.

SECONDARY OUTCOMES:
Determination of lymphocytic immune phenotypes in BAL and other biopsy samples by flowcytometry | 3 years
  To assess lymphocytic immune phenotypes in BAL and other biopsy samples from patients with IFI.
Measurement of cytotoxic T cell responses in blood samples from patients with IFI by ELISA | 3 years
  Assessment of T cell response on lymphocytes from peripheral blood
Correlation of survival at day 30 and 90 and immune checkpoint expression levels | 4 years
  To correlate the level of immune checkpoint expression with mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der Universität zu Köln, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellinghoff SC, Thelen M, Bruns C, Garcia-Marquez M, Hartmann P, Lammertz T, Lehmann J, Nowag A, Stemler J, Wennhold K, Cornely OA, von Bergwelt-Baildon MS, Schlosser HA. T-cells of invasive candidiasis patients show patterns of T-cell-exhaustion suggesting checkpoint blockade as treatment option. J Infect. 2022 Feb;84(2):237-247. doi: 10.1016/j.jinf.2021.12.009. Epub 2021 Dec 15. PMID 34921845